CLINICAL TRIAL: NCT06657469
Title: Effects of Computerized Progressive Attention Training Vs. Executive Functions Training in Children with ADHD
Brief Title: Computerized Attention Functions Training Vs. Executive Functions Training for Children with ADHD
Acronym: AFT-EFT-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Lilach Shalev, Prof., Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12123944
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Functions Training (AFT); Executive Functions Training (EFT); Neurocognitive Training; Cognitive Functions; ADHD Behavioral Symptoms
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — methylcobalamin-coenzyme M methyltransferase; Population Groups

STUDY DESIGN:
Intervention Model Description: In this study, participants were randomly assigned to one of three parallel groups: Attention Functions Training (AFT), Executive Functions Training (EFT), or a passive control group. Each group received a different intervention or no intervention, with the results being compared across groups to evaluate the relative effectiveness of each training program on attention, executive functions, academic performance, and behavior in children with ADHD.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and their parents were blinded to their group assignments within the intervention groups (AFT or EFT). However, participants and parents in the passive control group were aware of their assignment. Research assistants who conducted the assessments before, after, and at follow-up were blinded to all group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Attention Functions Training (AFT) Group (Experimental): The AFT group used two training tasks from the Cogmission software: A Conjunctive Continuous Performance Task (CCPT) designed to practice sustained attention, and a Go/No-go task, designed to practice response inhibition. This group also used three training tasks from the Computerized Progressive Attention Training (CPAT) program: (1) Conjunctive Visual Search Task, designed to improve selective-spatial attention; (2) Combined Orienting and Flanker Task, designed to improve orienting of attention; and, (3) Global-Local Task, designed to improve executive attention - conflict resolution. Each of the tasks consists of a broad hierarchy of difficulty levels, and the transition between them occurs after consistent improvement was obtained and performance reached a plateau at a given difficulty level.
  Interventions: Other: Attention Functions Training (AFT)
- Executive Functions Training (EFT) (Experimental): The EFT group used a computerized version of the Set game. Set is a pattern-recognition card game where players must identify sets of three cards that share or differ in specific attributes, such as color, shape, or number. It was used to train cognitive flexibility. In addition, this group used four computer games to train problem-solving. Three of them were designed by Leo De Sol Games and were based on familiar games: (1) Rush Hour; (2) Pipes/Plumber; and (3) Sliding Puzzle. The fourth game, Thinkrolls Kings & Queens by Avokiddo, is a challenging adventure puzzle game that incorporates logic and physics, requiring players to navigate mazes and overcome obstacles using reasoning. Additionally, three games developed by Mindware Consulting Inc. were used to train working memory based on well-known paradigms in the field.
  Interventions: Other: Executive Functions Training (EFT)
- Passive Control Group (No Intervention): Participants in this group did not receive any active intervention during the study period. They were assessed at the same time as the other groups-before the intervention and immediately after. This group enabled us to rule out spontaneous developmental effects, as well as learning and familiarity effects that may result from repeated exposure to the assessment tasks.

INTERVENTIONS:
Other: Attention Functions Training (AFT) — The AFT protocol included 18 group-based sessions, 75 minutes each, administered twice a week over a nine-week period. The training focused on improving sustained attention, selective-spatial attention, and executive attention through computerized tasks like the Conjunctive Continuous Performance Task and Go/No-Go tasks.
  Other Names: Attention Functions Training (AFT) Group
  Arms: Attention Functions Training (AFT) Group
Other: Executive Functions Training (EFT) — The EFT protocol included similar session structures with a focus on executive functions such as working memory, cognitive flexibility, and problem-solving. Tasks included computerized games such as visual puzzles.
  Arms: Executive Functions Training (EFT)

SUMMARY:
The goal of this clinical trial was to compare the effectiveness of two computerized neurocognitive training programs for children with Attention Deficit/Hyperactivity Disorder (ADHD) and to examine their impact on attention functions, executive functions, academic performance, and behavior. The main questions this study sought to answer were:

How does Attention Functions Training (AFT) compare to Executive Functions Training (EFT) in improving cognitive abilities related to attention and executive functions in children with ADHD? What are the effects of these programs on academic performance and behavior? Researchers compared the outcomes of the AFT group, the EFT group, and a passive control group, in order to determine which program was more effective across these domains.

Participants completed computerized training sessions focused on attention or executive functions twice a week for nine weeks. They also underwent cognitive, academic, and behavioral assessments at baseline, after the training, and at follow-up.

DETAILED DESCRIPTION:
This randomized controlled trial aimed to investigate and compare the effects of two distinct computerized neurocognitive training programs on children diagnosed with Attention Deficit/Hyperactivity Disorder (ADHD). The two interventions, Attention Functions Training (AFT) and Executive Functions Training (EFT), were designed to target different cognitive domains. The AFT program focused on improving sustained, selective-spatial, orienting, and executive attention, while the EFT program aimed at enhancing working memory, cognitive flexibility, and problem-solving abilities.

A total of 80 children with ADHD, aged 8-13 years, were randomly assigned to one of three groups: AFT, EFT, or a passive control group. Each training program included twice-weekly sessions over nine weeks. Participants underwent comprehensive assessments at three time points: baseline (pre-intervention), immediately after the intervention, and at a three-month follow-up. The assessments covered cognitive functions, academic skills, and behavioral symptoms as reported by parents.

The study employed repeated measures ANOVA to analyze the effects of the interventions. Primary outcome measures included improvements in attention and executive functions, with secondary measures focused on academic performance and parent-rated behavioral symptoms. Both short-term and long-term effects were assessed to evaluate the persistence of any observed improvements.

ELIGIBILITY:
Inclusion Criteria:

* ADHD

Exclusion Criteria:

* Coexisting diagnosis of other mental illness or neurological disorder (with the exception of ADHD and Learning Disabilities); previous serious head injury; uncorrected vision; additional developmental, sensory or motor issues; and if they are participating in other non-pharmacological treatment interventions specifically for ADHD (e.g., neurofeedback, cognitive-behavioral therapy, etc.).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-03-19 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
sustained attention | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  The CCPT (Conjunctive Continuous Performance Test ) was used to assess sustained attention. In this task, a series of geometric shapes of different colors were displayed on the monitor, and the participants were asked to press the spacebar each time the target stimulus (i.e., red square) appeared, and delay their responses when other stimuli, other than the target stimulus, were displayed. The task consisted of a single block of 320 trials, in which the target stimulus appears in only 30% of trials. Performance was measured by two important measures that are frequently used to evaluate sustained attention: (a) standard deviation of response times (SD of RT), calculated only for correct responses, which reflects inconsistency in RTs to targets; and (b) percentage of omission errors - in which the participant did not respond to the target stimulus. High values in these measures indicate a difficulty in sustained attention.
sustained attention | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  The Go/No-go Task. was also used to assess sustained attention. The task is similar to the CCPT except that the target stimulus appears in 70% of the trials (see Figure 3b for a schematic diagram of the task). Performance was measured by the same measures as the CCPT: (a) SD of RT; and (b) omission error rate.
selective-spatial attention | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  Conjunctive Visual Search Task (CVST). This task was designed to assess selective-spatial attention. In this task participants were asked to search for a blue square that appeared among an equal number of red squares and blue circles. There were four display sizes of 4, 8, 16 or 32 items, which were equally frequent and randomly intermixed within four 40-trial blocks. Participants were required to respond with their right index finger to the presence of the target and with their left index finger to its absence. RTs and accuracy rates were recorded for each display size with and without a target.
executive attention - conflict resolution | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  We used a Location-Direction Stroop-like Task (LDST) to assess executive attention - conflict resolution. The participants were instructed to make two types of judgment that referred to either the location or the direction of an arrow appearing on the screen. This arrow appears either above or below a fixation point and points upward or downward. On the first sub-task the participants were asked to respond only to the location of the arrow, while ignoring the arrow's direction. In the second sub-task the participants were asked to respond only to the direction of the arrow, while ignoring its location. Responses in both sub-tasks were the same - participants were directed to respond ''up'' with their right index finger and ''down'' with their left index finger. Each sub-task was comprised of two 40-trials blocks. Half of the trials within each block were congruent (e.g., an arrow located above the fixation point and directed upward) and half were incongruent.
problem solving | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  A computerized version ofTower of Hanoi Puzzle was used to evaluate problem solving ability. In this task, three pegs, numbered 1 to 3, appeared on the screen. On one of the pegs, three disks were arranged according to their size (i.e., the largest disk at the bottom and the smallest disk on top). The participants were instructed to move the disks from a starting position peg to a final position peg as fast as possible and with the least number of moves as possible, while using a third peg for their disposal. They were also asked to abide by three rules: (a) only one disk can move from peg to peg in each move; (b) a larger disk cannot be placed on top of a smaller one; and (c) all three pegs must be used.
auditory working memory capacity | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  The task WISC-IV Digit Span Forward was used to evaluate auditory working memory capacity. In this task, the participants were required to listen to and repeat a sequence of numbers read aloud by the research assistant. The task starts with the sequence length of only two digits and gradually increases in length up to nine digits. Participants have two chances at each sequence length, and the next length sequence is read to them only if one of the sequences in the previous length was repeated correctly. The measure we used for this task is the summary score, computed as the longest sequence remembered, multiplied by the number of correct sequences.
manipulation verbal information | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  We used the WISC-IV Digit Span Backward to evaluate the ability to manipulate verbal information while in temporary storage, namely, working memory's Central Executive. This task is very similar to the WISC-IV digit span forward, accept for two differences: (a) participants are asked to repeat the digits' sequence in the reversed order; and (b) the longest sequence is of eight digits.
visuospatial working memory capacity | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  We used a computerized version of the Corsi-Block Tapping Task Forward, to evaluate visuospatial working memory capacity. In this task, the participants were presented with a screen of 9 blocks. The blocks light up in a pre-fixed sequence, and the participants were instructed to click the blocks on the screen, using the computer mouse at the same order they were lit. The task starts with the sequence length of only two blocks and gradually increases in length up to nine blocks. Participants have two chances at each sequence length, and the next sequence length starts only if one of the sequences in the length before was repeated correctly.
  We also used Corsi-Block Tapping Task Backward to evaluate visuospatial working memory capacity. The task is very similar to the Corsi-Block Tapping Task Forward accept for two differences: (a) participants are asked to click on the blocks in the reversed order of their original presentation; and (b) the longest sequence is of eight blocks.
Fluid Intelligence | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  Fluid intelligence was evaluated by using the Raven's Colored Progressive Matrices. This test is designed for young children aged 5-11 years old, and consists of 36 items in three sets (A, AB, B), with 12 items per set. The three sets are arranged to assess the cognitive processes of which children under 12 years of age are usually capable of. The Raven's CPM produces a single raw score that can be converted to a percentile based on normative data.
Arithmetic | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  Arithmetic Task was comprised out of 40 arithmetic exercises that require utilizing the four basic operations: 20 exercises requiring adding and subtracting up to 20, and 20 exercises requiring multiplying and dividing up to a 100, intermixed. Participants were asked to solve as quickly and accurately as possible all exercises. Two measures were calculated out of this task: (a) speed - total time to finish the task (in sec); and (b) accuracy - the percentage of correct answers out of 40. The task was developed specifically according to the needs of this research.
Text Reading | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  Participants were asked to read aloud as fast and as accurate as possible, a Hebrew text that does not include syntactic movement. Prior to the administration of the task, the research assistant ensured the participants that they would not be asked questions regarding the content of the text, nor would they need to remember details from it. The research assistant recorded the participants' reading, documented their mistakes, and timed them. The main measures that were calculated for this task are: (a) the number of words read per minute (i.e., speed); and (b) the percentage of words read correctly.
Writing from Dictation | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  The research assistant dictated to the participants a text in Hebrew that included homophonic and pseudo-homophonic words. The participants were asked to write what was dictated to them as fast and as accurate as possible on a loose-leaf line paper. Two measures were calculated out of this task: (a) the number of words written per minute (i.e. speed); and (b) the percentage of words written correctly from all written words (i.e., accuracy).
Behavioral, Emotional and Social Performance | Baseline, post-intervention, follow-up (approximately 3 months after intervention)
  Parents completed three questionnaires online via Qualtrics:
  1. Attention Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV). 18 items rated on a 4-point scale (0 = never/rarely, 3 = very often).
     Range: 0 to 54, with higher scores indicating more severe ADHD symptoms.
  2. Child Behavior Checklist (CBCL). 113 items assessing 8 behavior syndromes. Range: depends on subscale, with higher scores indicating more problematic behaviors.
  3. Behavior Rating Inventory of Executive Function (BRIEF). 86 items assessing executive function on 8 subscales. Range: depends on subscale, with higher scores indicating more dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Lilach Shalev, Prof., Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
All de-identified participant data will be shared.
Time Frame: Data will be available upon request starting 6 months after the publication of the study results and will remain accessible for 5 years.
Access Criteria: Access to the de-identified participant data will be granted to researchers upon request. Researchers must provide a valid research proposal, including a clear study purpose and a plan for data use. Proposals must be approved by an Institutional Review Board (IRB) or an equivalent ethics committee. Access will be provided through a secure data-sharing platform upon approval.